CLINICAL TRIAL: NCT00923312
Title: Safety and Efficacy Phase I/IIa Trial of an RNActive®-Derived Cancer Vaccine in Stage IIIB/IV Non Small Cell Lung Cancer (NSCLC)
Brief Title: Trial of an RNActive®-Derived Cancer Vaccine in Stage IIIB/IV Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-9201-003
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2013-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CV9201 (Experimental): CV9201 is composed of five formulated mRNAs (drug product components) encoding antigens that are overexpressed or exclusively expressed in NSCLC cells.
  Interventions: Biological: CV9201

INTERVENTIONS:
Biological: CV9201 — CV9201 is a vaccine consisting of five drug product components. Treatment will be administered on 5 timepoints.

SUMMARY:
This is a phase I/IIa open, uncontrolled, international, prospective clinical trial, in an out-patient setting, in patients with stage IIIB/IV NSCLC.

The phase I part of the study consists of a dose escalation phase, in which the recommended dose (RD) for the phase IIa part of the study will be established based on the incidence of dose-limiting toxicities (DLT). In the phase IIa part of the study, additional patients will be included at the RD, to confirm the safety and explore the activity of that dose.

This study will take place in Switzerland (2 sites) and Germany (11 sites).

DETAILED DESCRIPTION:
Medical Need:

Lung cancer is the leading cause of cancer mortality in developed countries; about 87% of lung cancers are of the NSCLC type. Patients with more advanced but non-metastatic disease (IIIA or IIIB) usually undergo chemotherapy and/or radiation therapy, with or without secondary surgical resection. Patients with progression after chemotherapy and/or radiotherapy may receive second-line treatment with targeted therapies. Despite these aggressive treatments, only about 5% of patients with metastatic disease survive for 5 or more years. Given these dismal statistics, it is clear that new therapeutic approaches for treatment of NSCLC are urgently needed.

Potential Benefits:

CV9201 is an mRNA-based vaccine for the treatment of human NSCLC that is based on CureVac's RNActive® technology.

As an mRNA-based vaccine, CV9201 features several advantages over other approaches: it is highly specific, there is no restriction to the patient's MHC genotype, and it does not need to cross the nuclear membrane to be active. Finally, in the absence of reverse transcriptase, RNA can not be integrated into the genome.

For the planned first-in-man study, CV9201 will be administered in 5 doses. The phase I part of this phase I/IIa study is a dose finding study, to determine the RD for the phase IIa part.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and age ≥ 18 yrs and ≤ 75
2. Histologically or cytologically confirmed and documented stage IIIB /IV NSCLC
3. Documented stable disease or objective response according to RECIST criteria after initial chemotherapy or chemo-radiotherapy for advanced, unresectable disease:

   * Patients must have received a minimum of two cycles of standard chemotherapy, and adequate and effective radiotherapy if used in conjunction with chemotherapy (sequentially or concomitantly). Prophylactic brain radiation is allowed.
   * Surgery, radiotherapy and/ or chemotherapy can have been previously administered for non-advanced disease.
   * All therapies must be completed 4 weeks before start of study treatment.
4. Performance status: Eastern Cooperative Oncology Group (ECOG) 0 - 1
5. Life expectancy > 6 months as assessed by the investigator
6. Adequate organ function:

   * Bone marrow function: hemoglobin ≥ 100 g/L; white blood cell count (WBC) ≥ 3.0 x 109/L; lymphocyte count ≥ 1.0 x 109/L; absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelet count ≥ 100 x 109/L
   * Hepatic: aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times upper limit of normal (ULN) (≤ 5 x ULN if hepatic metastases present); bilirubin ≤ 1.5 x ULN
   * Renal: Creatinine ≤ 2 mg/ dL and creatinine clearance ≥ 45 mL/ min
7. Patients of child-producing potential must agree to use contraception while enrolled in the study and for one month after the last immunization
8. Written informed consent must be obtained prior to conducting any study-specific procedures.

Exclusion Criteria:

1. History of anti-cancer therapy for advanced disease other than initial chemotherapy or chemo-radiotherapy or surgery
2. Immunotherapy within 4 weeks prior to study enrollment, including cytokines such as G-CSF, GM-CSF or interferons
3. Treatment with investigational anti-cancer agents during initial therapy for advanced disease or any investigational agents within 4 weeks prior to study enrollment
4. Concurrent anti-tumor therapy or concurrent immunotherapy such as lectins, unspecific immunostimulants, etc.
5. Previous anti-cancer immunotherapy comprising RNA-transfected dendritic cells or DNA vaccines targeting any tumor-associated antigens
6. Concurrent systemic steroids except topical (inhaled, topical, nasal) for the last 28 days, except replacement therapy
7. Concurrent major surgery or planned surgery
8. Prior splenectomy
9. Documented history of active autoimmune disorders requiring systemic immunosuppressive therapy, (e.g., sarcoidosis, lupus erythematosus, rheumatoid arthritis, glomerulonephritis or systemic vasculitis), excepting autoimmune thyroiditis with only thyroid hormone replacement and stable disease > 1 year
10. Primary or secondary immune deficiency
11. Active allergy requiring continuous medication or active infections requiring anti-infectious therapy
12. Seropositive for HIV, HBV or HCV
13. History of other malignancies over the last 5 years (except basal cell carcinoma of the skin or carcinoma in situ of the cervix)
14. Uncontrolled medical condition considered as high risk for the treatment with an investigational drug including unstable diabetes mellitus, vena-cava-syndrome, known ascites and/or uncontrolled pleural effusion.
15. Brain metastases (symptomatic or asymptomatic) or leptomeningeal involvement
16. Symptomatic congestive heart failure (NYHA 3 and 4); unstable angina pectoris within 6 months prior to enrollment; significant cardiac arrhythmia, history of stroke or transient ischemic attack
17. History of seizures, encephalitis or multiple sclerosis
18. Gastric ulcer or inflammatory bowel disease or Crohn's disease or ulcerative colitis; no active diverticulitis
19. Active drug abuse or chronic alcoholism
20. Patients being committed to an institution by virtue of an order issued either by the judicial or the administrative authorities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-05; Primary Completion 2012-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Phase I: Determination of the recommended dose (RD) for exploration in the phase IIa part of the study | During the first 2-3 month of Phase I
Phase II: Assessment of safety and tolerability of the treatment regimen | Complete duration of Phase II

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Knuth, Prof. Dr., Principal Investigator — Universitätsspital Zürich
Locations (14):
- Germany (12):
  - RWTH Aachen, Aachen
  - Medizinische Klinik III, Universitätsklinikum Bonn, Bonn
  - Medizinische Klinik V, Klinikum Darmstadt, Darmstadt
  - Medizinische Klinik I, Universitätsklinikum Dresden, Dresden
  - Nordwest Krankenhaus, Frankfurt
  - Krankenhaus Großhansdorf, Großhansdorf
  - Universitätsklinikum Hamburg Eppendorf, Medizinische Klinik II, Hamburg
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - III. Medizinische Klinik und Poliklinik, Universitätsmedizin Mainz, Mainz
  - III. Medizinische Klinik, Klinikum rechts der Isar, München
  - Medizinische Klinik II, Universität Tübingen, Tübingen
- Switzerland (2):
  - UniversitätsSpital Basel, Basel
  - UniversitätsSpital Zürich, Zurich

REFERENCES:
- [Derived] Fotin-Mleczek M, Duchardt KM, Lorenz C, Pfeiffer R, Ojkic-Zrna S, Probst J, Kallen KJ. Messenger RNA-based vaccines with dual activity induce balanced TLR-7 dependent adaptive immune responses and provide antitumor activity. J Immunother. 2011 Jan;34(1):1-15. doi: 10.1097/CJI.0b013e3181f7dbe8. PMID 21150709
- See also: Homepage Sponsor — http://www.curevac.com